CLINICAL TRIAL: NCT04023084
Title: PDE4A Expression as a Biomarker of Responsiveness to Eucrisa
Brief Title: Response of Children With Atopic Dermatitis (Eczema) to Eucrisa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Anna Fishbein, MD, Attending Physician, Allergy & Immunology, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-2879
Record Dates: First submitted 2019-07-11; First posted 2019-07-17 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: dermatologic agents; surveys; questionnaires; topical therapy
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — crisaborole

STUDY DESIGN:
Intervention Model Description: children diagnosed with AD and aged 4 months-17 years old will receive intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atopic Dermatitis Group (Experimental): Receive crisaborole intervention
  Interventions: Drug: Crisaborole

INTERVENTIONS:
Drug: Crisaborole — Crisaborole 2% topical ointment applied twice daily to affected area(s) for 28 days
  Other Names: Eucrisa

SUMMARY:
The purpose of this study is to develop biomarkers to predict what medication is best for each child with atopic dermatitis (eczema). Participants will come in to Lurie Children's Allergy of Dermatology clinic for a skin examination and complete surveys. They will apply Eucrisa medication to their skin for 28 days before returning for a second and final skin examination and complete surveys. During these skin exams, tape will be placed on the skin and removed to collect skin cell samples. Photos will also be taken of the skin where tape was placed. There is an optional blood draw.

DETAILED DESCRIPTION:
The overall study design is an intervention open-label non-randomized clinical trial of Eucrisa treatment (Eucrisa is an FDA approved drug for this indication and in this age group) twice daily for 28 days in 5-17 year old children. This study intends to enroll 30 total participants. The main purpose of this study is to develop biomarkers to predict responsiveness to Eucrisa. The hypothesis that PDE4A is a strong driver of inflammation in atopic dermatitis (AD) patients with high PDE4A skin expression, and that they will be highly responsive to Eucrisa.

Based on a previously published study to use minimally invasive tape strip biomarkers to differentiate patient groups, a 30-fold difference was noted when comparing PDE4A expression levels between TH2 high and TH2 low patients (total n=30). The investigators anticipate that ~50% of patients will be responders per the primary outcome of improvement in clinician assessed disease severity (Investigator Global Assessment of Investigator's Static Global Assessment (ISGA)) defined as clear (0) or almost clear (1) with a 2-grade or more improvement from baseline. With a total sample size of 30, the investigators estimate ~15 will be responders and ~15 non-responders, with alpha=0.05, power=0.8, assuming standard deviation of log(2) to log(5) in mRNA expression difference. This would give power to see a difference in fold expression in the range of 1.9-4.1, and adequate power to see expected differences in the chosen biomarkers. Assuming 80% power, the investigators are also powered for secondary analyses to see correlations with biomarkers and secondary outcomes, with a correlation coefficient ≥ 0.5.

The investigators will recruit directly from the various clinics of Ann & Robert H. Lurie Children's Hospital (LC). Patients will be contacted for screening over the phone 2 weeks prior to their clinic visit and recruited in clinic for study participation.

If participants give permission over the phone, study staff will meet them when they come in for their Allergy or Dermatology clinic visit. On Days 1 (baseline visit) and 28 (final visit), the following procedures will be done. Their skin will be examined by a clinician, and transepidermal water loss (TEWL) will be measured using the non-invasive AquaFlux instrument. Skin samples will be taken from the participant's antecubital fossa and photographs will be taken only of the collection site via the tape stripping protocol. The samples will be stored without identifiers, only with the participant's study identification (ID) number. Photos will be stored on a password-protected computer, accessible only by study staff, without any identifiers and will be coded with study ID. Participants and their caregivers will also be asked to fill out questionnaires, including Patient-Reported Outcomes Measurement Information System (PROMIS) itch forms, PROMIS sleep items, and PROMIS Profile 25. The child will additionally complete a Patient-Oriented Eczema Measure (POEM) and a Children's Dermatology Life Quality Index (CDLQI). Parent and child will also complete daily diary entries regarding the child's Eucrisa application and will include a 10-point pruritus scale. All of these forms will be administered electronically, and the collected data will be maintained in a secure REDCap database. The electronic forms are set up such that participants must answer every item to complete the study. If they do not feel comfortable answering certain items, they may choose to discontinue involvement in the study without consequence. If, at the baseline visit only, the participant is already having blood drawn for another clinical indication, blood will additionally be drawn with their consent for study purposes (15 mL) for later RNA sequencing. Plasma and peripheral blood mononuclear cells (PBMCs) drawn at the initial visit in this subset of patients, will be frozen and stored (de-identified, in a locked freezer) at -80°C for later processing and correlation with tape strip biomarkers. The correct method of therapy application will be reviewed with the patient and/or caregiver. They will be advised to discontinue Eucrisa and seek medical attention immediately if signs or symptoms of hypersensitivity occur and to contact the study doctor. The research team will submit incident reports regarding adverse events to the Lurie Children's Institutional Review Board (IRB) via their Cayuse system. Subject ID numbers will be maintained separately from the data set. Source documents and case report forms are kept in a secured area (in a locked cabinet in a locked room) in the Department of Allergy & Immunology at Lurie Children's, and all electronic data is password-protected and will not be transmitted outside the Lurie server.

After isolating expression of putative biomarkers, specifically PDE4A. Primary analysis will compare baseline mean expression levels of PDE4A in "responder" versus "non-responder" groups. This will be defined by the primary clinical outcome of disease severity improvement by clinician assessment. The investigators anticipate data with a normal distribution, so a t-test will compare significance of average expression levels. If data is not normally distributed, comparisons will be made using the Mann-Whitney U test. Secondary analyses will look at mean differences between other biomarkers (TH2 (IL13, IL4R, CCL26), TH17/22 (IL36G), itch (ENKUR), and epidermal genes (FLG, LOR and S100A9) in the "responder" versus "non-responder" groups. In exploratory analyses, the investigators will evaluate whether these biomarkers changed while on Eucrisa at the 4 week follow up. Specifically, a paired samples t-test will be used (or Wilcoxon signed-rank test if data not normally distributed). Magnitude of change in biomarkers will also be descriptively compared to magnitude of clinical improvement in disease, similar to previously published methods.

To correlate quality of life measures at baseline with PDE4A expression levels, initially data will be graphed to visually inspect the distribution and association, with PDE4A expression on the X-axis and quality of life measures on the Y-axis. Pearson correlation coefficient will be used to evaluate the strength of the association, if non-normally distributed data, a Spearman correlation coefficient will be used to test associations. In exploratory analyses, the investigators will look at the relationship of these genes after treatment with PDE4A. Further analyses will be conducted to determine if patients will be categorized as responders or non-responders on all measures tested using clinically important differences in the tested measures. The investigators will compare responses to quality of life measures using descriptive statistics. Additionally, the investigators will also consider average PDE4A levels in responders versus non-responders using these assessment measures.

The investigators will also attempt to develop a logistic regression model to predict Eucrisa responders. Specifically, the investigators will look at the association between each biomarker and the outcome of interest. If significant, the investigators will include in the final model to determine the key biomarkers predicting Eucrisa responders.

The Lurie Children's IRB and will ensure that the research complies with all applicable policies and regulations through their Post-Approval Monitoring program. Their staff will review study documents, schedule and perform site visits with the investigators, and follow up with the research team on any findings to take the appropriate actions, if any.

ELIGIBILITY:
Inclusion Criteria:

* AD diagnosis by dermatologist or allergist based on Hanifin and Rajka criteria
* 5% or more treatable body surface area involvement
* baseline Investigator's Static Assessment (ISGA) score of mild (2) or moderate (3)
* patient on stable regimens (consistent use 14 days before day 1 of enrollment) of inhaled corticosteroids and antihistamines
* must have lesional skin in the antecubital fossa

Exclusion Criteria:

* use of topical corticosteroid, calcineurin inhibitor, or PDE4 inhibitor within 14 days of enrollment
* significant active infection
* any previous use of biologic therapy
* no pruritus at baseline visit, or other pruritic condition
* washing/moisturizer use 24 hours prior to tape strip biomarker collection at site
* uncontrolled asthma, uncontrolled allergic rhinitis, or other sleep disturbing condition

Ages: 4 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Changes in expression levels of biomarkers in responder versus non responder groups | Baseline (Day 1) and Day 28
  The baseline mean expression levels of biomarkers extracted from tape strips (TH2 (IL13, IL4R, CCL26), TH17/22 (IL36G), itch (ENKUR), epidermal genes (FLG, LOR and S100A9) and PDE4A will be compared in clinical "responder" versus "non-responder" groups. Groups will be defined by the primary clinical outcome of disease severity improvement by clinician assessment. Clinicians will assess disease severity by Investigator's Static Global Assessment (ISGA) and Eczema Area and Severity Index (EASI) score.

SECONDARY OUTCOMES:
Changes in Quality of life (anxiety, depressive symptoms, fatigue, mobility, pain interference, peer relationships) as assessed by PROMIS Pediatric Profile 25 and Correlation of changes with clinical responsiveness and biomarker PDE4A expression levels | Baseline (Day 1) and Day 28
  Changes in quality of life will be measured by comparing standardized PROMIS T-scores for each domain at Day 28 with baseline. The PROMIS Pediatric Profile 25 is a 25-item questionnaire and assesses anxiety, depressive symptoms, fatigue, mobility, pain interference, and peer relationships. Each item has five response options. The HealthMeasures Scoring Service will be used to calculate T-scores for each domain. A T-score of 50 is the average for the United States general population with a standard deviation of 10. A higher T-score represents more of the concept being measured. Responsiveness will be determined by comparing clinician-assessed disease severity by ISGA and EASI scores at baseline and Day 28.
Changes in Quality of life (symptoms and feelings, leisure, school or holidays, personal relationships, sleep, treatment) as assessed by CDLQI and Correlation of Quality of life changes with clinical responsiveness and biomarker PDE4A expression levels | Baseline (Day 1) and Day 28
  Changes in quality of life will be measured by comparing CDLQI scores at Day 28 with baseline. The CDLQI is a 10-item questionnaire assessing symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and treatment. Scores range from 0 to 30 and are calculated by summing the scores of each question. The higher the score, the more impaired quality of life. Responsiveness will be determined by comparing ISGA and EASI scores at baseline and Day 28.
Correlation of TEWL with clinical responsiveness and biomarker PDE4A expression levels | Baseline (Day 1) and Day 28
  Diffusion of water through the skin is measured using the AquaFlux instrument. Responsiveness will be determined by comparing ISGA and EASI scores at baseline and Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fishbein, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available after primary publication is accepted.
Access Criteria: Individual participant data will be publicly available through journal publication.

REFERENCES:
- [Background] Dyjack N, Goleva E, Rios C, Kim BE, Bin L, Taylor P, Bronchick C, Hall CF, Richers BN, Seibold MA, Leung DYM. Minimally invasive skin tape strip RNA sequencing identifies novel characteristics of the type 2-high atopic dermatitis disease endotype. J Allergy Clin Immunol. 2018 Apr;141(4):1298-1309. doi: 10.1016/j.jaci.2017.10.046. Epub 2018 Jan 6. PMID 29309794
- [Background] Paller AS, Tom WL, Lebwohl MG, Blumenthal RL, Boguniewicz M, Call RS, Eichenfield LF, Forsha DW, Rees WC, Simpson EL, Spellman MC, Stein Gold LF, Zaenglein AL, Hughes MH, Zane LT, Hebert AA. Efficacy and safety of crisaborole ointment, a novel, nonsteroidal phosphodiesterase 4 (PDE4) inhibitor for the topical treatment of atopic dermatitis (AD) in children and adults. J Am Acad Dermatol. 2016 Sep;75(3):494-503.e6. doi: 10.1016/j.jaad.2016.05.046. Epub 2016 Jul 11. PMID 27417017
- [Background] Paton DM. Crisaborole: Phosphodiesterase inhibitor for treatment of atopic dermatitis. Drugs Today (Barc). 2017 Apr;53(4):239-245. doi: 10.1358/dot.2017.53.4.2604174. PMID 28492291
- [Background] Hamilton JD, Suarez-Farinas M, Dhingra N, Cardinale I, Li X, Kostic A, Ming JE, Radin AR, Krueger JG, Graham N, Yancopoulos GD, Pirozzi G, Guttman-Yassky E. Dupilumab improves the molecular signature in skin of patients with moderate-to-severe atopic dermatitis. J Allergy Clin Immunol. 2014 Dec;134(6):1293-1300. doi: 10.1016/j.jaci.2014.10.013. PMID 25482871
- [Background] Simpson EL, Paller AS, Boguniewicz M, Eichenfield LF, Feldman SR, Silverberg JI, Chamlin SL, Zane LT. Crisaborole Ointment Improves Quality of Life of Patients with Mild to Moderate Atopic Dermatitis and Their Families. Dermatol Ther (Heidelb). 2018 Dec;8(4):605-619. doi: 10.1007/s13555-018-0263-0. Epub 2018 Oct 22. PMID 30345457
- [Background] Chamlin SL, Mattson CL, Frieden IJ, Williams ML, Mancini AJ, Cella D, Chren MM. The price of pruritus: sleep disturbance and cosleeping in atopic dermatitis. Arch Pediatr Adolesc Med. 2005 Aug;159(8):745-50. doi: 10.1001/archpedi.159.8.745. PMID 16061782